CLINICAL TRIAL: NCT00771173
Title: THE CAT(H) STUDY CATHETER ANALGESIA TRIAL Phenazopyrdine vs. Placebo: a Randomized Controlled Trial A CREST 2010 Project
Brief Title: CATHETER ANALGESIA TRIAL Phenazopyrdine vs. Placebo: a Randomized Controlled Trial
Acronym: CATH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Linda Brubaker, Professor of Medicine and Dean and Chief Diversity Officer, Stritch School of Medicine, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201073
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Catheter-related Bladder Discomfort
Keywords: Phenazopyrdine; post operative bladder catheritization; VAS scores; Bladder pain related to indwelling foley catheters.; Bladder irritaion related to indwelling foley catheters.
MeSH Terms: interventions — Phenazopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Medication Group (Active Comparator): Participants that are randomized to the phenazopyridine HCl group will receive the study medication (200 mg of phenzopyridine HCl orally) after leaving the operating room. We anticipate the first dose to be given after the patient has left the recovery area. We will continue use of study medication until it has been given up to 24 hours after the first VAS collection or catheter removal, whichever occurs first
  Interventions: Drug: phenazopyridine HCl
- Placebo tablet Group (Placebo Comparator): For participants randomized to the placebo group will follow the same dosing schedule for the study medication, although they will receive an inert placebo tablet.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: phenazopyridine HCl — Phenazopyrdine HCl 200 mg q8h x 24
  Other Names: Pyridium
  Arms: Study Medication Group
Other: Placebo — Placebo tablet administered q8 hours for 24 hours postop.
  Arms: Placebo tablet Group

SUMMARY:
The primary aim of this randomized clinical trial is to compare the utility of phenazopyridine HCl vs. placebo in reducing catheter-associated discomfort during the post-operative period in the gynecologic patient using mean VAS measurments.

DETAILED DESCRIPTION:
This is a randomized clinical trial to determine whether phenazopyridine HCl reduces catheter-related bladder discomfort, using mean VAS scores and overall pain medicine requirements in women catheterized following in-patient gynecologic surgery.

Hypothesis and Aims:

We plan to test the null hypothesis that there is no difference in post-operative pain as measured by VAS pain scores and pain medication requirements in women with a Foley catheter following gynecologic surgery that are given phenazopyridine HCl vs. placebo.

The primary aim of this randomized clinical trial is to compare the utility of phenazopyridine HCl vs. placebo in reducing catheter-associated discomfort during the post-operative period in the gynecologic patient using mean VAS measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women undergoing gynecologic surgery who are expected to tolerate oral medication within 12 post-operative hours and require an indwelling catheter for a minimum of 12 post operative hours after start of oral medication.

Exclusion Criteria:

1. Hypersensitivity to phenazopyridine products (Defined as a having a previous anaphylaxis reaction to phenazopyridine products).
2. Known contraindications to phenazopyridine HCl:

   * Renal failure or insufficiency (Defined as having abnormal renal function on previous laboratory testing (BUN/Cr) or as having a known renal disease).
   * History of hepatic disease or failure (Defined as having known liver disease or having elevated LFTs on previous laboratory testing. Patients who would not otherwise have such testing are not required to undergo special study labs).
   * Known glucose-6-phosphate dehydrogenase deficiency.
3. Simultaneous suprapubic catheterization.
4. Inability to take oral medication within 12 hours after surgery.
5. Pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Brubaker, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola Univeristy Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anderson C, Chimhanda M, Sloan J, Galloway S, Sinacore J, Brubaker L. Phenazopyridine does not improve catheter discomfort following gynecologic surgery. Am J Obstet Gynecol. 2011 Mar;204(3):267.e1-3. doi: 10.1016/j.ajog.2010.12.045. PMID 21376167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from September 2008 through December 2009 at the 2 Loyola system hospitals.
Pre-assignment Details: All enrolled patients were randomized to a group. Those patients who were enrolled but not included in statistical analysis was due to inconsistent collection of our primary outcome data. Nursing staff and house staff failed to collect VAS scores consistently.
Groups:
- Placebo Group: For participants randomized to the placebo group will follow the same dosing schedule for the study medication, although they will receive an inert placebo tablet.
  Blinding: The research pharmacist has facilitated the blinding by placing the active agent (200 mg tablets) into a solid colored capsule. She will make matching placebo capsules filled with lactose powder. To aid in blinding and avoid systemic administration of other dye agents for women in the placebo group, a small amount of orange dye will be placed in the Foley bag. This has been tested in the planning for this trial and is known effectively color the urine orange.
- Active Agent Group: Participants that are randomized to the phenazopyridine HCl group will receive the study medication (200 mg of phenzopyridine HCl orally) after leaving the operating room. We anticipate the first dose to be given after the patient has left the recovery area. We will continue use of study medication until it has been given up to 24 hours after the first VAS collection or catheter removal, whichever occurs first
Period: Overall Study
Arm/Group | Placebo Group | Active Agent Group
Started | 129 | 129
Completed | 107 | 112
Not Completed | 22 | 17

BASELINE CHARACTERISTICS:
Groups:
- Active Agent Group: Participants that are randomized to the phenazopyridine HCl group will receive the study medication (200 mg of phenzopyridine HCl orally) after leaving the operating room. We anticipate the first dose to be given after the patient has left the recovery area. We will continue use of study medication until it has been given up to 24 hours after the first VAS collection or catheter removal, whichever occurs first
  phenazopyridine HCl: Phenazopyrdine HCl 200 mg q8h x 24
- Placebo Group: For participants randomized to the placebo group will follow the same dosing schedule for the study medication, although they will receive an inert placebo tablet.
  Placebo: Placebo tablet administered q8 hours for 24 hours postop.
- Total: Total of all reporting groups
Arm/Group | Active Agent Group | Placebo Group | Total
Number analyzed (Participants) | 129 | 129 | 258
Age, Continuous [Mean (Full Range); unit: years] | 54 [40 to 75] | 53 [40 to 75] | 54 [40 to 75]
Sex/Gender, Customized [Number; unit: participants]
  Women | 129 | 129 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 126 | 129 | 255
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 105 | 103 | 208
  More than one race | 5 | 8 | 13
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Catheter-associated Discomfort During the Post-operative Period in the Gynecologic Patient Using Mean Visual Analogue Scale (VAS) Measurments
Description: The VAS measures bladder pain on a straight line from 0 to 10 in centimeters, where a mark of zero indicates no pain and a mark of 10 indicates worst possible pain. Mean VAS score was recorded for participants in the active treatment and placebo cohorts.
Time Frame: 24 hours
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Active Agent Group | Placebo Group
Number analyzed (Participants) | 112 | 107
centimeters | 0.95 (1.8) | 0.97 (1.7)
Statistical Analysis 1: Comparison: Active Agent Group vs Placebo Group; The independent samples t-test was used to test the null hypothesis that the mean VAS score for the active treatment cohort (i.e., those receiving pyridium) was no different than the mean VAS score for those receiving placebo; Test type: Superiority or Other; p = .745, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were recorded over the course of 24 hours during participants' hospitalization.
Arm/Group | Active Agent Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/107
Other Adverse Events (participants affected / at risk) | 0/112 | 0/107

LIMITATIONS AND CAVEATS:
One limitation of our study was inconsistent collection of our primary outcome data. Nursing staff and house staff failed to collect VAS scores consistently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No